CLINICAL TRIAL: NCT04574232
Title: SporTRIA Study: A Multicentre Trial for Excretion Kinetics of Triamcinolone Acetonide Following Sport Related Intra-articular Injections in Knees; Definitions of the Washout Periods
Acronym: SporTRIA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Edem ALLADO, Doctor, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2020-A01448-31
Record Dates: First submitted 2020-09-18; First posted 2020-10-05 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Doping in Sport; Glucocorticoids
Keywords: glucocordicoids; Doping; sport; urinary
MeSH Terms: interventions — Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- athletic subjects (Other): athletic subjects who may need intra-articular knee infiltration
  Interventions: Drug: knee intra-articular infiltration with Triamcinolone acetonide

INTERVENTIONS:
Drug: knee intra-articular infiltration with Triamcinolone acetonide — knee intra-articular intra-articular ultrasound-guided infiltration of Triamcinolone acetonide

SUMMARY:
Intra-articular and peri-articular glucocorticoid (GC) injections are common in sports medicine. However, from 1st January 2022, all injectable GC routes (including intra-articular administration (IA)) will be prohibited in-competition by World Anti-Doping Agency (WADA). Due to these rules, an IA GC treatment out-of-competition could result in an adverse analytical finding (AAF) in-competition if the washout period is not clearly defined. The aim of this study is to determine the urinary excretion profile of triamcinolone acetonide following IA to help in the definition of the washout periods.

ELIGIBILITY:
Inclusion Criteria:

* Sports practice at least 4h / week
* No comorbidities against indicating intra-articular knee injection
* Subject with a knee disease requiring intra-articular injection of GCs

Exclusion Criteria:

* Subject with glucocorticoid (GC) allergy or GC medical contraindication
* Pregnant women or women of childbearing potential without effective contraception
* Washout period of all injectable routes and systemic use of GCs less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Determination of the excretion profile of triamcinolone acetonide in urine following intra-articular ultrasound-guided injection | Change from baseline, pre-injection (day 0) to date (up to 35 days) where glucocorticoids urinary value below the 15 ng/ml
  For subjects with a glucocorticoids urinary value below the 15 ng/ml threshold at D0 (before injection), identification of the date (up to 35 days) following the intra-articular ultrasound-guided injection which will correspond in the standards of the World Agency (under 15 ng/ml)

SECONDARY OUTCOMES:
Modeling of the excretion profile of triamcinolone acetonide in urine following intra-articular ultrasound-guided injection. | evolution glucocorticoids urinary value from baseline, pre-injection (day 0) to Day 35
  Evolution of urinary triamcinolone acetonide concentration
Determination of the excretion profile of cortisol in urine following intra-articular ultrasound-guided injection to evaluate systemic effect | Change from baseline, pre-injection (day 0) glucocorticoids urinary value up to 35 days
Determination of the excretion profile of triamcinolone acetonide in DBS anti-doping test following intra-articular ultrasound-guided injection. | Change from baseline, pre-injection (day 0) glucocorticoids DBS value up to 35 days
Modeling of the excretion profile of triamcinolone acetonide in DBS anti-doping test following intra-articular ultrasound-guided injection. | evolution glucocorticoids blood value from baseline, pre-injection (day 0) to Day 35
  Evolution of blood triamcinolone acetonide concentration
Determination of cortisol levels in DBS to evaluate systemic effect | Change from baseline, pre-injection (day 0) glucocorticoids DBS value up to 35 days
Identification of GCs on hair mark presence one month after intra-articular ultrasound-guided injection of triamcinolone acetonide. | Change from baseline, pre-injection (day 0) glucocorticoids hair value up to 35 days
Evaluation of the impact of exogenous corticosteroids on endogenous steroids profile (androgens and GCs) in DBS samples. | Change from baseline, pre-injection (day 0) glucocorticoids DBS value up to 35 days
  Mesure of blood exogenous corticosteroids on endogenous steroidsconcentration

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Régional Universitaire de Nancy., Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: Yes
The data from all patients will be centrally stored in Nancy. Data management will be carried out by CHRU de Nancy (Direction de la Recherche et de l'Innovation). The conditions for data transfer of all or part of the study database are decided by the study sponsor and are the subject of a written contract. This study and the data collected fall within the scope of Reference Methodology MR001.
  The data may be transmitted to the companies in the group to which the promoter belongs and to its contractual partners in a form which should not permit the direct or indirect identification of persons lending themselves to research

REFERENCES:
- [Derived] Allado E, Poussel M, Gambier N, Saunier V, Starck M, Buisson C, Cinquetti G, Albuisson E, Chenuel B. SporTRIA study-a multicentre trial protocol for excretion kinetics of triamcinolone acetonide following sport-related intra-articular injections in knees: definitions of the washout periods. BMJ Open. 2021 Jun 9;11(6):e047548. doi: 10.1136/bmjopen-2020-047548. PMID 34108168